Effect of Monazite Sands in Patients with Osteoarthritis of the Knee Ethical committee Protocol No: 3.160.891

Meeting\_minutes\_template

## TEMPLATE FOR MINUTES OF MEETING

| Summary | | | | | | |
|---|---|---|---|---|---|---|
| Meeting Topic | | | | | | |
| Date | | From | To | | | |
| Location | | Note Taker | | Duration | | |
| Study brief Title: Effects of Sand Treatment on Osteoarthritis | | | | | | |
| Official Title: Effect of Monazite Sands in Patients with Osteoarthritis of the Knee | | | | | | |
| Ethical committee Protocol No: 3.160.891 Unique Protocol ID: T015-M02-2019AF002 | | | | | | |
| Agenda | | | | | | |
| Tin | me Topic | | | | | |
| | Attendee List | | | _ | _ | |
| # | Name | | - | Present | Reason | n of Absence |
| 1 | | | | | | |
| 2 | | | | | | |
| Meeting Notes | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| Action Items | | | | | | |
| # | Task | | Person Responsible | | | <b>Due Date</b> |
| 1 | | | | | | |
| 2 | | | | | | |
| Prepared By: | | | | | | |
| Dat | | | | | | |
| | viewed By: | | | | | |
| | Date | | | | | |

